CLINICAL TRIAL: NCT02307188
Title: Atrial Signal Analysis Using a Multipolar Catheter in Patients Undergoing Atrial Fibrillation and Flutter Ablations
Brief Title: Multipolar Mapping and Atrial Arrhythmias
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Angelo Biviano (Other)
Responsible Party: Sponsor-Investigator, Angelo Biviano, Associate Professor of Medicine, Columbia University
Organization: Columbia University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: AAAN3357
Record Dates: First submitted 2014-11-25; First posted 2014-12-04 (Estimated); Results first posted 2016-03-16 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2016-02

CONDITIONS: Atrial Fibrillation or Atrial Flutter
Keywords: Atrial Fibrillation; Atrial Flutter; Multipolar Catheter; Atrial Arrhythmia
MeSH Terms: conditions — Atrial Fibrillation; Atrial Flutter

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Basket Catheter (Experimental): The Constellation Full Contact Mapping Catheter (multipolar catheter) to be utilized for collection of atrial electrograms.
  Interventions: Device: Constellation Full Contact Mapping Catheter

INTERVENTIONS:
Device: Constellation Full Contact Mapping Catheter — 64-electrode intracardiac mapping catheter.

SUMMARY:
This clinical investigation utilizes the Constellation Full Contact Mapping catheter in the left and right atria to explore atrial signal characteristics that can guide atrial fibrillation and atrial flutter ablation procedures more effectively.

DETAILED DESCRIPTION:
Atrial fibrillation (AF) and atrial flutter (AFL) are the most common cardiac arrhythmias in adults, and account for a substantial portion of patient morbidity and healthcare expenditures. Great effort has been put forth to discover effective treatments for AF/FL. Promising results of catheter ablation suggest that AF/FL may be eliminated in a majority of patients. For example, data from numerous laboratories shows that up to 85 percent of patients with the paroxysmal form of AF may be free of recurrences and off anti-arrhythmic drugs at one year follow-up.

ELIGIBILITY:
Inclusion Criteria:

Patients referred to the PI (Dr. Biviano) or co-investigators in the Program of Cardiac Electrophysiology at Columbia University Medical Center who are scheduled to undergo ablation will be approached for recruitment:

* Older than 45 years of age
* History of AF and/or AFL and are candidates for catheter ablation.

Exclusion Criteria:

Patients not fitting the above clinical criteria or unwilling to comply with the instructions of the monitor are excluded, as well as patients with the following:

* Permanent leads or prosthetic or stenotic valves present
* Active systemic infection
* Echocardiographically-confirmed visual presence of thrombus
* For whom the inability of obtaining vascular access exists
* Heparin-induced thrombocytopenia
* Hemodynamic instability or shock

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2014-11; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Angelo B Biviano, MD, MPH, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Five (5) patients were enrolled. The catheters were used in the left atrium in one (1) patient. The remaining patients were excluded because of subtherapeutic activated clotting time levels < 300 seconds (3 patients) or presence of prosthetic valve (1 patient).
Groups:
- Basket Catheter: The Constellation Full Contact Mapping Catheter (multipolar catheter) to be utilized for collection of atrial electrograms.
  Constellation Full Contact Mapping Catheter: 64-electrode intracardiac mapping catheter.
  Since enrollment began, a total of five (5) patients consented to enrollment in the study during their atrial fibrillation/tachycardia ablation procedures. The catheter (a new catheter was used for each patient) was used in the left atrium in one patient who met all inclusion criteria and did not have any exclusions.
Period: Overall Study
Arm/Group | Basket Catheter
Started | 5
Completed | 1 (Four of 5 patients did not meet required criteria to complete the study after they were enrolled.)
Not Completed | 4

BASELINE CHARACTERISTICS:
Population: Due to the paucity and lack of quality of intracardiac electrogram information collected from the one patient for whom the catheter was used in the left atrium, the collected electrogram data were not analyzed further.
Arm/Group | Basket Catheter
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Atrial Fibrillation Dominant Frequency
Description: Electrogram signal analysis will be performed to assess the dominant frequency of the atrial fibrillation electrograms collected by this catheter. These values will be correlated to patient outcomes.
Time Frame: 1 year
Population: Because the quality of intracardiac electrogram data for the one patient to complete the study was not sufficient for analysis, this outcome measure was not analyzed.
Groups:
- Basket Catheter: The Constellation Full Contact Mapping Catheter (multipolar catheter) to be utilized for collection of atrial electrograms.
  Constellation Full Contact Mapping Catheter: 64-electrode intracardiac mapping catheter.
  Five (5) patients were enrolled. The catheters were used in the left atrium in one (1) patient. The remaining patients were excluded because of subtherapeutic ACT levels < 300 seconds (3 patients) or presence of prosthetic valve (1 patient).
  Due to the paucity of information collected from the one patient for whom the catheter was used in the left atrium, the collected electrogram data were not analyzed further.
Arm/Group | Basket Catheter
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Potential adverse events were collected at time of catheter insertion up to 1 day after procedure.
Groups:
- Basket Catheter: The Constellation Full Contact Mapping Catheter (multipolar catheter) to be utilized for collection of atrial electrograms.
  Constellation Full Contact Mapping Catheter: 64-electrode intracardiac mapping catheter.
  No adverse events related to this catheter were noted.
Arm/Group | Basket Catheter
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No